CLINICAL TRIAL: NCT03347591
Title: Rare Bleeding Disorders in the Netherlands
Acronym: RBIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Academisch Ziekenhuis Maastricht (Other); Erasmus Medical Center (Other); Maxima Medical Center (Other); Academisch Ziekenhuis Groningen (Other); UMC Utrecht (Other); Leiden University Medical Center (Other); Haga Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HEMSTOL47
Record Dates: First submitted 2017-10-25; First posted 2017-11-20 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Rare Bleeding Disorders
Keywords: Fibrinogen; Factor II; Factor V; Factor V & VIII; Factor VII; Factor X; Factor XI; Factor XIII; α2-antiplasmin; Plasminogen activator inhibitor 1; Epidemiology; Genetics; Phenotype
MeSH Terms: interventions — Hemostasis; Fibrinolysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with rare bleeding disorders: All patients registered in Dutch Haemophilia Treatment Centers with known disorders of the coagulation factors fibrinogen, factor II, V, V & VIII, VII, X, XI, XIII, α2-antiplasmin and plasminogen activator inhibitor type 1, aged 1 years and older.
  Interventions: Genetic: WES; Diagnostic Test: Several assays

INTERVENTIONS:
Genetic: WES — 136 bleeding related OMIM (Online Mendelian Inheritance in Man)-proved genes involved in haemostasis will be selected from Whole Exome Sequencing (WES)
Diagnostic Test: Several assays — Patients will be approached by their own treating physician. Data will be collected through questionnaires, a clinical interview, a blood and saliva sample obtained from each participant, and thorough review of electronic patient records. All procedures are study related. In case a physician visit with the treating physician is already planned, or in case a venepuncture for regular diagnostics or treatment is already planned, this can be combined with the study procedures to prevent an extra visit.
  Other Names: Hemostasis (several screening tests, several diagnostic tests, global assay); Fibrinolysis; Lupus anticoagulans; Anti β2 glycoprotein

SUMMARY:
Rationale: Rare bleeding disorders (deficiency of fibrinogen, factor II, V, V&VIII, VII, X, XI, XIII, α2-antiplasmin or plasminogen activator inhibitor 1) are not well defined with respect to their clinical phenotype, laboratory phenotype en genotype. At present, little is known about their clinical presentation, bleeding scores, bleeding episodes, health-related quality of life, laboratory parameters, genetics and current treatment. There are large differences in bleeding tendency and weak correlations with the level of factor deficiencies. Therefore, it is essential to perform thorough research in patients with rare bleeding disorders and perform laboratory and genetic tests, to seek explanations for the variety in clinical phenotype.

Objective: The purpose of the RBIN study is to describe the epidemiology, bleeding tendency, laboratory parameters, quality of life and genetics of all known patients in the Netherlands with rare bleeding disorders. In addition, the study aims to examine the relationship between clinical phenotype, laboratory phenotype and genotype.

Study design: explorative cross-sectional multicenter observational study Study population: all patients registered in Dutch Haemophilia Treatment Centers with known disorders of the coagulation factors fibrinogen, factor II, V, V & VIII, VII, X, XI, XIII, α2-antiplasmin and plasminogen activator inhibitor type 1, aged 1 years and older.

Main study parameters/endpoints:

Description of the clinical phenotype, laboratory phenotype, genotype and quality of life.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: participating patients will be invited for one visit to their treatment center in order to draw blood, take a saliva sample and perform questionnaires. This will take approximately 40 to 120 minutes. Since the population of patients with rare bleeding disorders is very small it is important to include all patients, also minors (children <18 years), in the study (around one third of known patients are minors). Therefore, this study may be regarded as group-related. The risk associated with participation is negligible.

DETAILED DESCRIPTION:
Primary objectives:

* Describe the epidemiology, clinical presentation, bleeding score, bleeding episodes, quality of life, laboratory parameters, genetics and treatment of homozygous and known heterozygous individuals (of all ages) with rare bleeding disorders (disorders of fibrinogen, FII, FV, FV & VIII, FVII, FX, FXI, FXIII, alpha-2-antiplasmin and PAI-1 deficiency) in the Netherlands;
* Examine the relationship between the clinical and laboratory presentation (clinical and laboratory phenotype), and between phenotypes and genetics (genotype);
* Examine the relationship between quality of life, phenotype and genotype;
* Validate the established factor activity levels for patients to remain without symptoms.

Secondary objectives:

* Compare the clinical presentation, bleeding score, quality of life and laboratory parameters of individuals with a rare bleeding disorder (disorders of fibrinogen, FII, FV, FV & VIII, FVII, FX, FXI, FXIII, alpha-2-antiplasmin and PAI-1 deficiency) to those of individuals with haemophilia A or B in cooperation with the HIN-6 investigators
* Establish a firm base for a future Dutch registry for homozygous and known heterozygous individuals with rare bleeding disorders
* To develop a standard set of patient-reported, clinical and administrative data to be collected on a regular basis
* Liaise with the pro-RBDD study, a similar study in Italy, to work towards a pan-European study linking phenotype to genotype in individuals with rare bleeding disorders
* To assess if the NHA can distinguish mild clinical phenotypes in patients with similar factor activity levels
* To evaluate the usefulness of saliva coagulation biomarker tests in the management of patients with a rare bleeding disorder
* To examine whether age-dependent laboratory changes in factor concentrations and fibrinolysis occur in individuals with rare bleeding disorders and if so, whether they influence clinical phenotype
* To evaluate if patients with rare bleeding disorders are protected from arterial thrombosis

ELIGIBILITY:
Inclusion Criteria:

* Established homozygous or known heterozygous rare bleeding disorder due to deficiency or dysfunction of fibrin, FII, FV, FV & FVIII, FVII, FX, FXI, FXIII, alpha-2-antiplasmin and PAI-1 ;
* Age 1 year and older;
* For patients ≥ 16 years old; written informed consent.
* For patients 12-16 years old; written informed consent from both the patient and their parents/legal guardian(s).
* For patients <12 years old; written informed consent from their parents/legal guardian(s).

Exclusion Criteria:

* No informed consent given;
* Residency outside of the Netherlands

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: To date, 394 patients with a rare bleeding disorder are known to the eight Dutch centers that treat such patients. Approximately one third of these patients are homozygous; and around two thirds are heterozygous individuals.
  All known homozygous and heterozygous patients with a rare bleeding disorder will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-11-07 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Epidemiology | 1 year
  Determine the prevalence of rare bleeding disorders in the Netherlands by evaluating all patients known in all Dutch Haemophilia Treatment Centers
Phenotype | 1 year
  Clinical phenotype will be measured by bleeding scores measured as ISTH-BAT.
Laboratory phenotype | 1 year
  Measure the factor concentrations of all patients known with a Rare Bleeding Disorder in the Netherlands
Quality of Life | 2 years
  Quality of life will be measured using the RAND-36 questionnaire
Genotype | 2 years
  Determine the genotype of patients (homozygous, heterozygous, compound heterozygous) by whole exome sequencing

SECONDARY OUTCOMES:
Minimum factor level | 1 year
  The minimum factor level necessary to remain without bleeding will be calculated by measuring factor levels in all patients and their bleeding scores by ISTH-BAT
Age | 1 Year
  To examine whether age-dependent laboratory changes in factor concentrations and fibrinolysis occur in individuals with rare bleeding disorders and if so, whether they influence clinical phenotype.

CONTACTS AND LOCATIONS:
Overall Officials: S. Schols, PhD, Principal Investigator — Radboud University Medical Center
Locations (7):
- Netherlands (7):
  - Academisch Medisch Centrum, Amsterdam
  - Maxima Medisch Centrum, Eindhoven
  - University Medical Center Groningen (UMCG), Groningen
  - Maatricht UMC+, Maastricht
  - Radboud university medical center, Nijmegen
  - Erasmus MC, Rotterdam
  - Haga hospital, The Hague

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Derived] Saes JL, Verhagen MJA, Meijer K, Cnossen MH, Schutgens REG, Peters M, Nieuwenhuizen L, van der Meer FJM, Kruis IC, van Heerde WL, Schols SEM. Bleeding severity in patients with rare bleeding disorders: real-life data from the RBiN study. Blood Adv. 2020 Oct 27;4(20):5025-5034. doi: 10.1182/bloodadvances.2020002740. PMID 33064819

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03347591/Prot_SAP_000.pdf